CLINICAL TRIAL: NCT06179836
Title: Chinese Severe Brain Injury Trial
Acronym: CSBIT
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: CSBIT
Record Dates: First submitted 2023-12-10; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Severe Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good prognosis group
- poor prognosis group

SUMMARY:
Building a Large Chinese Cohort(Chinese Severe brain injury Trial）

ELIGIBILITY:
Inclusion Criteria:

* a clear cause of brain injury
* disorders of consciousness, GCS≤12
* within six months of onset

Exclusion Criteria:

* not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with impaired consciousness with a clear cause of brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale | 6 months after severe Brain Injury
  The unabbreviated scale title is Glasgow Outcome Scale. GOS includes a score of 1-5, with the higher the score, the better the prognosis.

SECONDARY OUTCOMES:
Glasgow Outcome Scale | 3 months and 12 months after severe Brain Injury
  The unabbreviated scale title is Glasgow Outcome Scale. GOS includes a score of 1-5, with the higher the score, the better the prognosis.

IPD SHARING:
Plan to Share IPD: No